CLINICAL TRIAL: NCT06172673
Title: A Database for Emotion Analysis Using Physiological and Psychological Assessment by 40FY
Status: Completed | Type: Observational
Sponsor: 40FY (Industry)
Responsible Party: Sponsor
Other Study IDs: DEAP-40FY
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Psychological Stress; Heart Rate Variability; Mental Health Services
Keywords: Contactless measurement of Heart Rate Variability; Mobile digital mental health monitoring; Psychological assessment
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Community dwelling participants: Individuals between the ages of 19 and 45 in South Korea.

SUMMARY:
A comprehensive study examining the physiological, emotional and psychological aspects of stress among Korean adults

DETAILED DESCRIPTION:
A dataset for the analysis of affective states of Korean adults. Participants' facial and finger videos were recorded using a cell phone camera, while watching six emotion-eliciting video stimuli, each three minutes in length (two of each: neutral, positive, and negative). Participants were asked to rate their emotion and arousal in terms of arousal and valence levels. The ECG data were collected using a 1-lead ECG while watching the six emotion-eliciting video stimuli. Psychological assessments were conducted using self-administered scales measuring psychological status and personality.

ELIGIBILITY:
Inclusion Criteria:

* Adults over the age of 19 and under the age of 45.

Exclusion Criteria:

* Participants vulnerable to voluntary consent, such as those who have evidence of intellectual disability or traumatic brain injury
* Participants who have difficulty reading and understanding Korean.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: We recruited Adults between the ages of 19 and 45 who can read fluently in Korean. All study participants understood the study procedures and provided written informed consent according to the Declaration of Helsinki.
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2023-07-19 (Actual); Primary Completion 2023-12-08 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale (PSS) | Baseline
  The PSS is a 10-item scale that measures the perceived stress on a 5-point severity with higher scores indicating more severe perceived stress.
Center for Epidemiologic Studies Depression Scale (CES-D) | Baseline
  The CES-D is a 20-item questionnaire that measures depressive symptoms on a 4-point likert scale.
State-Trait Anxiety Inventory (STAI) | Baseline
  The STAI is a 40-item inventory that measures state and trait anxiety. Higher score means higher anxiety.
Beck Anxiety Inventory (BAI) | Baseline
  A 21-item self-inventory on a 4-point likert scale measuring common somatic and cognitive symptoms of anxiety.
Five Factor Model of Personality Short Form Test (IPIP-NEO-120) | Baseline
  The five factor model of personality is the most widely accepted and used personality based on trait theory. IPIP-NEO-120 has been developed to reduce the number of questions to 120 while maintaining the structure of 30 sub-facets comprising 5 factors of the 300-item. The shortened version has been reported to have high validity and reliability.
Schema Scale | Baseline
  A 35-item questionnaire developed by 40FY for identifying 5-types of maladaptive schema types. The questionnaire consists of 5-point Likert scale. The Schema Scale was developed based on schema theory and other psychodynamic theories. The scale was developed by a certified psychiatrist and 3 clinical psychologists. A higher score for each factor means that the individual has more severe maladaptive psychological schemas.
Depression, Anxiety, and Stress Scale (DASS-21) | Baseline
  The DASS-21 scale is an abbreviated version of the 42-item DASS test to measure depression, anxiety, and stress. It consists of seven items for each domain and is rated on a 4-point Likert scale.
Screening for Anxiety Disorders in Adults (SCAARED) | Baseline, Follow-up
  A 44-item, 3-point Likert scale, self-report questionnaire developed as a screening test for anxiety disorders in the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5). Items from the Screen for Children Anxiety Related Disorders (SCARED) was adapted for the adult version and validated a appropriate for screening for anxiety disorders.
Self-Assessment Manikin Scale (SAM) | Baseline
  The SAM consists of five pictures, with reference points between the pictures, which are rated on a 9-point scale. Participants are asked to mark their emotion and arousal on the picture closest to their emotional state. Six emotion-eliciting video stimuli (2 neutral, 2 negative, and 2 positive) are given, and individuals rate emotion and arousal right after watching each video stimuli.
Heart-rate variability indices (SDNN, RMSSD, LF, HF) | Baseline
  Measured from 1-lead ECG device. SDNN is the standard deviation of the NN interval. It is an indicator of the stability of the cardiovascular system and the responsiveness of the heart rhythm. RMSSD is the root mean square value of the variation of consecutive NN intervals, which indicates the activity of mainly parasympathetic nerves. The ECG data were collected by 1-lead ECG while watching 6 emotion-eliciting video stimuli.

CONTACTS AND LOCATIONS:
Overall Officials: Woori Moon, MD, PhD, Principal Investigator — 40FY, Inc.
Locations (1):
- Research and Development Division, 40FY Inc., Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No